CLINICAL TRIAL: NCT04820088
Title: Simulated Conversation Training for Mental Healthcare Providers to Improve Care for Transgender and Gender Nonconforming Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SIMmersion, LLC (Industry)
Collaborators: Towson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Improving Care Delivery
Record Dates: First submitted 2021-03-04; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Gender Affirming Communication Skills
Keywords: Communication Skills; Gender
MeSH Terms: conditions — Coitus | interventions — Glutamyl Aminopeptidase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The educational intervention will be TTACS, the training program with simulated roleplays. Each participant will be asked to schedule 10 hours of time to utilize the simulation. In order to ensure all participants adhere to the minimum intervention requirements, each will be asked to schedule training time with a member of the research team. Participants will attend an initial training session where each participant will receive a short orientation about the product and its capabilities. Participants will attend an initial training session at one of two sites Psychology Department at Towson University or SIMmersion's office in Columbia, MD based on participant preference. Subsequent training sessions may be completed at Towson, SIMmersion or can be completed individually. Participants will receive confirmation emails the day before a scheduled session and a phone call to reschedule any missed sessions.
  Interventions: Other: Computer based role play trianing
- Contro Arm (No Intervention): Students randomized to the control group will be given an electronic copy of the Guidelines for Psychological Practice with Transgender and Gender Non-Conforming People (APA, 2015) and asked to take notes in the pdf document. The amount of time students spend on the document and note-taking will be recorded and notes will be analyzed for content. As an incentive, the participants in the control group will be given access to TTACS after they complete the post-intervention assessment.

INTERVENTIONS:
Other: Computer based role play trianing — Participants will train with a computer-based role-play simulation. They will interact with a lifelike video character on screen. They will interact with the character in one of four scenarios (i.e., patient intake, traditional needs, high-risk needs,and social and physical transition). They will receive real-time and after-action feedback in a safe, non-stressful environment. Their usage of the system will be monitored and transcripts will be collected.
  Other Names: American Psychological Association Guidelines for Psychological Practice with Transgender and Gender Non-Conforming People (APA, 2015)
  Arms: Intervention Arm

SUMMARY:
Phase I: Eligible participants (n=20) will be recruited to participate in a feasibility evaluation of the client intake module to be developed. Participants will complete pre- and post-intervention knowledge assessment outcome measures. The gain score, defined as the difference between the pre-training and post-training score, will be calculated for each participant. Each participant will spend up to 2 hours interacting with the intervention. Additionally, an implementation focus group (n=6) of administrators, educators, and key decision-makers will be conducted to assess the feasibility of implementing the proposed training suite in their programs.

Phase II: During Phase II, participants (n=100) will complete in two standardized patient encounters pre- and post-intervention to evaluate the efficacy of the proposed training suite. Participants assigned to the intervention group will receive 10 hours of training with the product and will be asked to complete a Training Experience Questionnaire after their post-intervention standardized patient encounter. Control group participants will receive the APA guidelines for Psychological Practice with Transgender and Gender Non-Conforming People for review. Control group participants will submit their notes taken while reviewing the guidelines. It is expected that the intervention group will show increased knowledge, skill, awareness, and cultural competency when working with the target population as measured by the Standardized Patient encounters as rated on a Standardized Patient Checklist. Additionally, the team anticipates the experimental group participants will rate the training suite as easy to use, relevant, and realistic.

DETAILED DESCRIPTION:
Phase I:

In order to assess feasibility and measure success in development, the team will recruit 20 providers in training from multiple sites around the United States to utilize the Intake Module to determine if the product changes provider knowledge. SIMmersion and their collaborators successfully used this methodology in a prior SBIR Fast-Track proposal to train health care providers in suicide assessment skills (R44 MH114710).

Hypothesis: The investigative team hypothesizes that there will be a positive gain score on the knowledge assessment for a majority of the participants after interacting with the training simulation for one hour.

Outcome Data:

Demographics: Participants will complete a demographic questionnaire related to age, sex, race, ethnicity, area of licensure, years of experience, prior training experience and experience with TGNC populations.

Usage Data: Each participant will be asked to complete the simulated conversation within the module a minimum of two times. The program will automatically store their usage data.

Product Evaluation: Upon completion of the post-test knowledge assessment, participants will be asked to provide feedback related to the usefulness, feasibility, scalability, appropriateness, ability to practice, and engagement level of the simulation using Likert scales (0-10) and open-ended questions.

Phase II:

Control Group: Students randomized to the control group will be given an electronic copy of the Guidelines for Psychological Practice with Transgender and Gender Non-Conforming People (APA, 2015) and asked to take notes in the pdf document. The amount of time students spend on the document and note-taking will be recorded and notes will be analyzed for content. As an incentive, the participants in the control group will be given access to TTACS after they complete the post-intervention assessment.

Educational Intervention: The educational intervention will be TTACS, the training program with simulated roleplays. Each participant will be asked to schedule 10 hours of time to utilize the simulation. In order to ensure all participants adhere to the minimum intervention requirements, each will be asked to schedule training time with a member of the research team. Participants will attend an initial training session where each participant will receive a short orientation about the product and its capabilities. Participants will attend an initial training session at one of two sites Psychology Department at Towson University or SIMmersion's office in Columbia, MD based on participant preference. Subsequent training sessions may be completed at Towson, SIMmersion or can be completed individually. Participants will receive confirmation emails the day before a scheduled session and a phone call to reschedule any missed sessions.

While the program will be set up as a ready-to-use training package, prior research efforts have shown that requiring participants to utilize the training product in a computer lab provides consistent compliance rates which lead to a more accurate evaluation of the product's efficacy. However, given the demanding nature of practicing students' schedules, requiring all intervention usage at our two sites may be difficult for participants. The research team anticipates that the proposed method will accommodate for participant schedules while still ensuring intervention compliance.

Demographic Collection: All training participants will complete a questionnaire designed to gather background information on demographic characteristics and other important characteristics. Information collected will include age, gender, race, program enrollment, prior exposure/training in working with TGNC individuals, and current coursework. This data will permit between-group comparability during subsequent data analysis.

Performance Improvement Assessment Using Standardized Patient Methodology (H1-H4). The skills test will consist of two Standardized Patient (SP) testing stations, as described above. Each station is set up in 30-minute units. Prior to counseling each SP, participants will have 5 minutes to review scenario instructions. This will provide background information on the client's previous encounters with the clinician, if any. Then, the participant will have 25 minutes to work with the SP.

Ten SPs will be recruited and trained by the staff at Towson University and Dr. Mastroleo. Training will be conducted in 3-hour sessions and include scenario, demonstration role-plays and/or videotapes, observed script practice sessions, group discussion of the character they are portraying and the questions that may be asked. They will also be taught how to time and score (using the checklist) the sessions.Dr. Mastroleo has been training SPs for intervention trials for the past 10 years and is well equipped to do so for this project.

Methods to Ensure Reliability of Standardized Patient Performance: All SP interactions will be audio recorded for review and further evaluation. The research team will review the first 5 tapes of each SP and every 5th tape thereafter to ensure the SPs are following the script and scenario protocol. It is the researchers' experience that 10-20% of SPs are not able to follow the script despite extensive training. Utilizing this review methodology identifies these SPs immediately so they can be replaced with SPs that can adhere to the study protocols.

Training Experience Questionnaire: Upon completion of the post-intervention SP encounters, each participant in the intervention arm will be asked to complete a Training Experience Questionnaire (TEQ) which will allow them to evaluate TTACS using a series of 5-point Likert scale questions and open-ended prompts. The research team anticipates that participants will indicate agreement or strong agreement on the TEQ that the product is (H5) an acceptable training tool (i.e., easy-to-use, realistic, relevant) and contributes to their skill development.

ELIGIBILITY:
Phase I:

Feasibility Evaluation: Participants (n=20) will be masters and doctoral candidates from M.A. and Ph.D. psychology programs. Participants will meet the following inclusion criteria:

(1) Currently enrolled full-time in one of the following programs: The University of Massachusetts-Boston Clinical Ph.D. Program, the University of Kentucky M.A. and Ph.D. programs in Counseling Psychology, the University of Tennessee Ph.D. program in Counseling Psychology, and the Palo Alto University Ph.D. Program in Clinical Psychology (see letters of support).

Participants will be excluded for the following:

No participants will be excluded on the basis of race, gender, background, or ethnicity.

Implementation Focus Group (n=6):

Participants will be included if they are the director of a psychology program or provider training organization. Participants will be excluded if they have (1) uncorrected vision or hearing problems that prevent using the software. No participants will be excluded on the basis of race, gender, background, or ethnicity.

Phase II:

Randomized Controlled Trial (RCT):

In Phase II participants (n=100) in the Randomized Controlled Trial (RCT) are students enrolled in graduate clinical and counselling psychology programs in the Baltimore/Washington D.C. area. The study will include male and female subjects, all 18 years of age or older. One-Hundred (100) participants will be enrolled, from those that apply by a specified deadline, that meet the following inclusion criteria:

(1) Currently enrolled full-time in one of the following programs: Towson University Counseling M.A. Program, Towson University Clinical M.A. Program, Howard University Counseling Ph.D. program, and The George Washington University graduate program in LGBT Health (see letters of support).

Participants will be excluded if:

No participants will be excluded on the basis of race, gender, background, or ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-02 (Estimated); Study Completion 2021-10-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge Assessment | Phase I, Month 6
  The research team will create a bank of 45 multiple-choice questions related to Intake and general cultural competencies including, gender , and communication skills. These will align and correlated with the skills in the training program. The program will randomly select 20 questions for each participant's pre-test. For the post-test, the program will randomly select 20 of the remaining 45 questions to ensure that individual participants are not assesed with repeat questions. AS no evidence-based based knowledge assessment measure exists related to the targeted skills, the team will rely on the expertise of investigative team and expert consultants to create the question bank. These questions will be informed by minority stress theory, intersectionality theory and multicultural competency frameworks. To ensure that participants are not learning from the test, answers and total scores will not be revealed to participants.
Standardized Patient Checklist | Phase II, Months 17-22
  The team, with assistance from the expert panel, will create behavior checklists for each SP scenarios. These SP Checklists will be based on 15 items, using a yes/no/partial scoring format (i.e., the subject demonstrated the required skill); each item will be given 5 points (yes), 0 points (no), or 2 points (partial), respectively. There will be an additional 25 points awarded based on overall performance focused on empathy, rapport building, and general communication skills. The primary teaching objectives to be included on the checklists will be informed by APA Guidelines (2015) and identified by the team and converted into yes/no/partial question format. This methodology has proven successful in past SBIRs in which the SPs evaluated the participant after the encounter (i.e., R42-AA016486, R44-AA022265, R44-DP003845, R44-DA026229, and R44-MH080496).
Training Experience Questionnaire | Phase II, Months 17-22
  Upon completion of the Phase II intervention period and the Standardized Patient performance improvement assessment, each participant in the intervention arm will be asked to complete a Training Experience Questionnaire (TEQ) which will allow them to evaluate TTACS using a series of 5-point Likert scale questions and open-ended prompts.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - SIMmersion, Columbia, Maryland
  - Towson University, Towson, Maryland

IPD SHARING:
Plan to Share IPD: Undecided